CLINICAL TRIAL: NCT05161182
Title: Westlake Personalized Nutrition Intervention Study: N-of-1 Trials for Dietary Macronutrient Intake 2
Brief Title: Westlake N-of-1 Trials for Macronutrient Intake 2 ( WE-MACNUTR 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20211011ZJS001
Record Dates: First submitted 2021-11-18; First posted 2021-12-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-10

CONDITIONS: Postprandial Hyperglycemia; Metabolic Disorder, Glucose
Keywords: Personalized Nutrition; Glucose Metabolism; Gut Microbiota
MeSH Terms: conditions — Hyperglycemia; Glucose Metabolism Disorders | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat, low carbohydrate diet (Experimental)
  Interventions: Other: High fat, low carbohydrate diet
- Low fat, high carbohydrate diet (Experimental)
  Interventions: Other: Low fat, high carbohydrate diet

INTERVENTIONS:
Other: High fat, low carbohydrate diet — Throughout the 5-day intervention, participants are provided with a high fat, low carbohydrate (HF-LC) diet in which the percentage of fat, protein and carbohydrate is 60%, 15% and 25%, respectively.
  Other Names: HF-LC
  Arms: High fat, low carbohydrate diet
Other: Low fat, high carbohydrate diet — Throughout the 5-day intervention, participants are provided with a low fat, high carbohydrate (LF-HC) diet in which the percentage of fat, protein and carbohydrate is 10%, 15% and 75%, respectively.
  Other Names: LF-HC
  Arms: Low fat, high carbohydrate diet

SUMMARY:
Diet and nutrition are key to maintain human health. Westlake N-of-1 Trials for Macronutrient Intake (WE-MACNUTR) trial investigates individualized postprandial glycemic responses to different proportions of dietary fat and carbohydrates intake using an n-of-1 experimental study design. The experimental diets are isocaloric high fat, low carbohydrate (HF-LC) or low fat, high carbohydrate (LF-HC). With standardized intervention and strictly controlled eating behaviors, the WE-MACNUTR study identifies specific HC-responders and HF-responders in terms of postprandial glucose response.

This is a follow-up study offered to participants who have completed the WE-MACNUTR study in 2019. Volunteers will be asked to participate in four 5-d periods while wearing glucose monitors (Abbott Freestyle Libre) with the following experimental sequence: 1) a washout diet, 2) HF-LC or LC-HF diet, 3) a washout diet, 4) HF-LC or LC-HF diet. The experimental diet will be randomly assigned. Participants will be asked to provide a fasted blood sample and to collect fecal, urine and saliva samples at each visits.

DETAILED DESCRIPTION:
This study is a two arm dietary intervention study. Participants will be recruited from the WE-MACNUTR study based on the defined inclusion and exclusion criteria. The study duration will last up to 21 days.

Volunteers will be asked to participate in four 5-day periods while wearing glucose monitors (Abbott Freestyle Libre) with the following experimental sequence: 1) a washout diet, 2) HF-LC or LC-HF diet, 3) a washout diet, 4) HF-LC or LC-HF diet. The experimental diet will be randomly assigned.

Participants will enter the study on a usual (washout) diet and will have a 5-day run in period for baseline data collection. Participants will be asked to follow dietary guidance and consumed a healthy and balanced diet during this period.

ELIGIBILITY:
Inclusion Criteria:

* Participants have completed WE-MACNUTR trial in 2019
* Participants have no traveling plans within 1 months
* Participants are able and willing to comply with the study protocol and provide informed consent

Exclusion Criteria:

* Refuse or are unable to provide informed consent to participate in the study
* Have long-term gastrointestinal diseases and take daily relevant medications
* Have taken antibiotics in the last 2 weeks
* Have type 2 diabetes and are taking medications or other treatments
* Have chronic or acute liver disease and are taking medications or other treatments
* Have cardiovascular diseases and are taking medications or other treatments
* Have kidney disease and are taking medications
* Suffer from chronic anxiety or depression, or other critical neuronal disorder and/or history of relevant medication
* Are pregnant or lactating, or are planning to be pregnant in the next 3 months
* Diagnosed with an eating disorder (e.g. anorexia nervosa or bulimia nervosa)
* Are vegan, or unwilling to consume foods provided in the study
* Have history of alcohol or drug addiction, or smoke above 15 cigarettes per day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Blood glucose profiling | 20 days
  Real-time blood glucose fluctuations will be recorded by CGM.

OTHER OUTCOMES:
Urines untargeted metabolomics profiling | Day 6, day 11 day 16 and day 21 of the study
  Urine metabolite extracts will be analysed by performing liquid chromatography/quadrupole time-of-flight mass spectrometry (LC/Q-TOF/MS). Compound will be identified by retention time and relative amount.
Fecal targeted metabolomics profiling | Day 6, day 11 day 16 and day 21 of the study
  Fecal metabolite extracts will be analysed by performing liquid chromatography/quadrupole time-of-flight mass spectrometry (LC/Q-TOF/MS). Metabolites, L-alanine for example, will be identified in μmol/L.
Microbiome taxonomic profiling | Day 6, day 11 day 16 and day 21 of the study
  Stool samples will be collected on day 6, day 11 day 16 and day 21 of the study. Shotgun metagenomic sequencing will be performed in stool samples. The taxonomic profiling and the organisms' relative abundance will be quantified using MetaPhlAn.
Serum metabolomics profile | Day 6, day 11 day 16 and day 21 of the study
  Venous blood samples will be collected at fasting in the morning on day 6, day 11 day 16 and day 21 of the study. The liquid chromatography/mass spectrometry (LC/MS) method with targeted metabolomics will be performed in blood serum. Compound (amino acids, fatty acids and bile acids) will be identified by retention time and relative amount.
Lipid metabolism | Day 6, day 11 day 16 and day 21 of the study
  Triglyceride, cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, apolipoprotein A1 and apolipoprotein B will be analyzed at all visits of the study.
Body composition | Day 5 of the study
  Body composition (fat mass, lean mass in kg ) will be assessed by bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China